CLINICAL TRIAL: NCT04251585
Title: Single Center Safety and Tolerability Trial of Intranasal Insulin in Parkinson's Disease
Brief Title: Intranasal Insulin in Parkinson's Disease
Acronym: INI-PD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: HealthPartners Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: A19-214
Record Dates: First submitted 2020-01-28; First posted 2020-02-05 (Actual); Results first posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Parkinson Disease
Keywords: intranasal; insulin
MeSH Terms: conditions — Parkinson Disease; Insulin Resistance

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of 3 treatment groups or the placebo group.
  * 20 international units twice daily (n=7)
  * 40 international units twice daily (n=7)
  * 80 international units twice daily (n=9)
  * placebo (n=7)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All participants, care providers, investigators, and outcomes assessors are masked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Low Insulin (Experimental): Regular insulin (Novolin-R) 20 international units (10 units) in one nostril twice daily for 21 days, 100 µl volume.
  Interventions: Drug: Regular Novolin R
- Medium Insulin (Experimental): Regular insulin (Novolin-R) 40 international units (10 units) in each nostril twice daily for 21 days, 100 µl volume.
  Interventions: Drug: Regular Novolin R
- High Insulin (Experimental): Regular insulin (Novolin-R) 80 international units (10 units) in each nostril twice daily for 21 days, 200 µl volume.
  Interventions: Drug: Regular Novolin R
- Placebo (Placebo Comparator): 0.9% sodium chloride in each nostril twice daily for 21 days, 100 µl volume.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Regular Novolin R — Intranasal insulin
  Arms: High Insulin; Low Insulin; Medium Insulin
Drug: Placebo — Intranasal placebo (0.9% saline)
  Arms: Placebo

SUMMARY:
This project will investigate exploratory outcomes related to the effect of intranasal insulin on cognition, mood, apathy and motor performance of subjects with Parkinson's disease over a 3 week period.

DETAILED DESCRIPTION:
Parkinson's disease (PD) is the second most common neurodegenerative disease after Alzheimer's dementia and was originally described as a motor disease. The diagnosis of PD is still based on the core motor features of bradykinesia, resting tremor, and rigidity, primarily as a result of degeneration of nigrostriatal dopaminergic neurons. In addition to the classic motor symptoms, however, PD is increasingly recognized as a multisystem disorder. A variety of non-motor symptoms, including cognitive deficits and dementia, are commonly observed in patients with PD.

In this study, we aim to investigate which intranasal insulin dose out of three doses and placebo, administered at three different doses or placebo over a 21-day period, is the optimum dosage based on safety and tolerability in Parkinson's disease. A similar design was used in a trial investigating intranasal oxytocin in frontotemporal dementia. Dosing for the first two groups of this study is based on previously conducted intranasal insulin studies in Alzheimer's disease (AD) and mild cognitive impairment (MCI), using daily doses on 20 and 40 IU of intranasal insulin. Higher dose have been found to be safe in healthy adults. Prior studies performed have demonstrated favorable effects of this regimen in the MCI/AD population without peripheral hypoglycemia.

ELIGIBILITY:
Inclusion Criteria:

* Subject has Idiopathic PD defined by the cardinal sign, bradykinesia, plus the presence of at least 1 of the following: resting tremor or rigidity and without any other known or suspected cause of Parkinsonism (according to Movement disorder society (MDS) clinical diagnostic criteria for Parkinson's disease confirmed by a fellowship trained movements disorder specialist
* Subject is Hoehn & Yahr stage less than or equal to 3
* Subject has a MOCA score ≥10.
* Subject is > 40 and <90 years of age.
* Female subjects are post-menopausal or have a negative pregnancy test
* The subject must be proficient in speaking, reading and understanding English in order to comply with procedural testing of cognitive function, memory and physiology.
* Subject has provided informed written consent prior to participation. In the event that subject is legally unable to provide informed written consent due to deterioration in cognitive abilities, fully informed written consent must be provided by a legally authorized representative.
* Subject is on a stable dose (at least 1 month prior to baseline visit) of antiparkinsonian agents and is willing to remain on this dose for the duration of the study. If the subject is on a cholinesterase inhibitor, a stable dose without changes for 1 month is also required.
* Subject has undergone a brain CT or MRI prior to the study as part of their previous diagnostic workup for PD to rule out underlying structural lesions, as determined clinically significant by the investigator

Exclusion Criteria:

* Subject has atypical Parkinson's syndrome(s) due to drugs (e.g., metoclopramide, neuroleptics), metabolic neurogenetic disorders (e.g., Wilson's Disease), encephalitis, cerebrovascular disease, or degenerative disease (e.g., Progressive Supranuclear Palsy, Multiple System Atrophy, Corticobasal Degeneration, Lewy Body dementia)
* Subject has medical history and/or clinically determined disorders: chronic sinusitis, untreated thyroid disease, or significant head trauma.
* Subject has history of any of the following: moderate to severe pulmonary disease, poorly controlled congestive heart failure, significant cardiovascular and/or cerebrovascular events within previous 6 months, condition known to affect absorption, distribution, metabolism, or excretion of drugs such as any hepatic, renal or gastrointestinal disease or any other clinically relevant abnormality that inclusion would pose a safety risk to the subject as determined by investigator.
* Subject has had previous nasal and/or oto-pharyngeal surgery and severe deviated septum and/or other anomalies.
* Subject has history of any psychiatric illness that would pose a safety risk to the subject as determined by investigator.
* Subject is currently taking sedative medications that are clinically contraindicated as determined by investigator.
* Subject has undergone a recent change (<1 month) in their anti-parkinsonian medication, cholinesterase inhibitor or anti-depressant medication.
* Subject has current or recent drug or alcohol abuse or dependence as defined by Diagnostic and Statistical Manual of Mental Disorders, fourth edition, text revision (DSM-IV TR).
* Screening laboratory results that are medically relevant, in which inclusion would pose a safety risk to the subject as determined by investigator.
* Subject has participated in a clinical trial investigation within 3 months of this study.
* Subject has an insulin allergy.
* Subject has Insulin-dependent diabetes

Ages: 41 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2020-02-04 (Actual); Primary Completion 2024-08-27 (Actual); Study Completion 2024-08-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julia C Johnson, MD, Principal Investigator — HealthPartners Neurology
Locations (1):
- HealthPartners Neuroscience Center, Saint Paul, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One participant was deemed ineligible prior to randomization. One participant completed treatment but was removed before analysis following the revision of eligibility criteria around MOCA score. 28 participants who completed treatment and were eligible were included in the analysis.
Period: Overall Study
Arm/Group | Low Insulin | Medium Insulin | High Insulin | Placebo
Started | 6 | 7 | 10 | 6
Completed | 6 | 7 | 9 | 6
Not Completed | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Low Insulin | Medium Insulin | High Insulin | Placebo | Total
Number analyzed (Participants) | 6 | 7 | 9 | 6 | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.3 (5.0) | 63.4 (5.1) | 68.2 (4.9) | 69.2 (6.1) | 67.3 (5.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 5 | 4 | 16
  Male | 3 | 3 | 4 | 2 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 0 | 1
  Not Hispanic or Latino | 6 | 6 | 9 | 6 | 27
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 6 | 7 | 9 | 6 | 28
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Montreal Cognitive Assessment (MoCA) [Mean (Standard Deviation); unit: units on a scale] — The Montreal Cognitive Assessment (MoCA) is a widely used screening assessment for detecting cognitive impairment. Range: 0-30. Lower score indicates more cognitive impairment.
  units on a scale | 26.8 (1.8) | 27.3 (2.7) | 24.6 (3.0) | 24.5 (1.9) | 25.7 (2.7)
UPDRS [Mean (Standard Deviation); unit: units on a scale] — The unified Parkinson's disease rating scale (UPDRS) is used to follow the longitudinal course of Parkinson's disease. The UPD rating scale is the most commonly used scale in the clinical study of Parkinson's disease. Range: 0-260. Higher score indicates more disability from Parkinson's disease.
  units on a scale | 24.2 (13.8) | 24.5 (11.1) | 24.4 (12.0) | 24.3 (8.2) | 24.4 (10.8)
Baseline HbA1C [Mean (Standard Deviation); unit: percent] — A hemoglobin A1C (HbA1C) test is a blood test that shows average level of blood glucose, over the past two to three months. A higher level indicates more glucose in the blood.
  percent | 5.7 (.2) | 5.5 (.2) | 5.6 (.5) | 5.6 (.2) | 5.6 (.3)

OUTCOME MEASURES:

1. Primary Outcome: Safety Measured by Count of Safety Events
Description: Composite safety event - this is a count of either a reduction of fasting glucose to <70 mg/dL or an unintended reduction of weight >5%. A larger composite event count indicates a less safe treatment.
Time Frame: 3 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Low Insulin | Medium Insulin | High Insulin | Placebo
Number analyzed (Participants) | 6 | 7 | 9 | 6
Participants | 0 | 0 | 0 | 0

2. Primary Outcome: Safety Measured by Fasting Glucose
Description: Pre-post change in fasting glucose (mg/dL). A larger decrease in fasting glucose indicates a less safe treatment.
Time Frame: baseline and 3 weeks
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Low Insulin | Medium Insulin | High Insulin | Placebo
Number analyzed (Participants) | 6 | 7 | 9 | 6
mg/dL | -3.8 [-6.9 to -1.0] | -1.3 [-6.8 to 4.2] | -5.9 [-10 to -1.8] | -3.8 [-9.8 to 2.1]

3. Primary Outcome: Safety Measured by Body Weight
Description: Pre-post change in body weight (lbs). An unintended decrease in body weight indicates a less safe treatment.
Time Frame: baseline and 3 weeks
Measure: Mean (95% Confidence Interval); unit: pounds
Arm/Group | Low Insulin | Medium Insulin | High Insulin | Placebo
Number analyzed (Participants) | 6 | 7 | 9 | 6
pounds | -0.63 [-1.8 to 0.50] | 0.34 [-1.6 to 2.3] | -0.33 [-1.9 to 1.3] | -0.55 [-3.0 to 1.9]

4. Primary Outcome: Safety Measured by the Number of Serious Adverse Events (SAE) and Adverse Events (AE)
Description: Total number of AEs/SAEs during the course of treatment. More AEs/SAEs indicates a less safe treatment.
Time Frame: 3 weeks
Measure: Mean (Standard Deviation); unit: number of events
Arm/Group | Low Insulin | Medium Insulin | High Insulin | Placebo
Number analyzed (Participants) | 6 | 7 | 9 | 6
number of events
  SAE | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  AE | 2.8 (1.2) | 5.0 (2.8) | 2.0 (3.8) | 3.0 (0.89)

5. Secondary Outcome: Cognitive Function Measured by the Montreal Cognitive Assessment (MoCA)
Description: Pre-post difference. Total sum of scores. Range: 0-30. Higher score indicates less memory loss
Time Frame: 5 weeks
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Low Insulin | Medium Insulin | High Insulin | Placebo
Number analyzed (Participants) | 6 | 7 | 9 | 6
score on a scale | -1.0 [-3.0 to 1.0] | -0.71 [-2.5 to 1.1] | 0.67 [-0.93 to 2.3] | 0.5 [-1.5 to 2.5]

6. Secondary Outcome: Cognitive Function Measured by the Weschler Adult Intelligence Scale - Fourth Edition (WAIS-IV) Digit Span
Description: Pre-post difference. Scaled score. Range: 1-19. Forward and backward. Lower score indicates more impairment.
Time Frame: 3 weeks
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Low Insulin | Medium Insulin | High Insulin | Placebo
Number analyzed (Participants) | 6 | 7 | 9 | 3
score on a scale
  Forward Digit Span | 1.5 [-0.33 to 3.3] | 1.0 [-0.69 to 2.7] | 0.2 [-1.3 to 1.7] | 1.0 [-0.83 to 2.8]
  Backward Digit Span | 0.0 [-2.0 to 2.0] | -0.43 [-2.3 to 1.5] | 0.0 [-1.7 to 1.7] | 2.3 [0.29 to 4.4]

7. Secondary Outcome: Cognitive Function Measured by the Trailmaking Test Part A Time
Description: Pre-post difference. T-score. Mean: 50, Standard deviation: 10. A higher T-score indicates a better outcome/performance. Clinically, 1-1.5 standard deviations would be significant, 2 standard deviations would be considered abnormal/impaired.
Time Frame: baseline and 3 weeks
Measure: Mean (95% Confidence Interval); unit: T-score
Arm/Group | Low Insulin | Medium Insulin | High Insulin | Placebo
Number analyzed (Participants) | 6 | 7 | 9 | 6
T-score | 4.5 [-3.3 to 12.3] | 5.3 [-1.9 to 12.5] | 4.7 [-1.6 to 11.1] | 5.8 [-1.9 to 13.6]

8. Secondary Outcome: Cognitive Function Measured by the Trailmaking Test Part B Time
Description: as for outcome 7
Time Frame: baseline and 3 weeks
Measure: Mean (95% Confidence Interval); unit: T-score
Arm/Group | Low Insulin | Medium Insulin | High Insulin | Placebo
Number analyzed (Participants) | 6 | 7 | 9 | 6
T-score | 3.5 [-3 to 10] | 5.6 [-0.43 to 11.6] | 2.1 [-3.2 to 7.4] | -2.8 [-9.3 to 3.7]

9. Secondary Outcome: Cognitive Function Measured by the Trailmaking Test Parts A & B Errors
Description: Pre-post difference. Total number of errors. No range. More errors indicate more impairment.
Time Frame: 3 weeks
Measure: Mean (95% Confidence Interval); unit: number of errors
Arm/Group | Low Insulin | Medium Insulin | High Insulin | Placebo
Number analyzed (Participants) | 6 | 7 | 9 | 6
number of errors | 0 [-1.8 to 7.8] | 0 [-0.53 to 0.53] | -0.56 [-1.5 to 0.40] | 0 [-0.66 to 0.66]

10. Secondary Outcome: Cognitive Function Measured by the Judgement of Line Orientation
Description: Judgement of Line Orientation is an assessment of visuospatial ability. A Z-score of 0 represents the population mean. Pre-post difference. A positive difference indicates an improvement.
Time Frame: baseline and 3 weeks
Measure: Mean (95% Confidence Interval); unit: Z-score
Arm/Group | Low Insulin | Medium Insulin | High Insulin | Placebo
Number analyzed (Participants) | 6 | 7 | 9 | 6
Z-score | 0.06 [-0.64 to 0.70] | 0.19 [-0.38 to 0.77] | -0.44 [-0.94 to 0.07] | 0.21 [-0.41 to 0.84]

11. Secondary Outcome: Cognitive Function Measured by the Logical Memory Scaled Scores
Description: Pre-post difference. Scaled score. Range: 1-19. Logical memory immediate and delayed. Lower score indicates more impairment.
Time Frame: baseline and 3 weeks
Measure: Mean (95% Confidence Interval); unit: scaled score
Arm/Group | Low Insulin | Medium Insulin | High Insulin | Placebo
Number analyzed (Participants) | 6 | 7 | 9 | 6
scaled score
  Immediate Recall | 2.7 [0.23 to 5.1] | 2.4 [0.17 to 4.7] | 1.3 [-0.66 to 3.3] | 3.5 [1.1 to 5.9]
  Delayed Recall | 1.7 [-0.15 to 3.5] | 4.0 [2.3 to 5.7] | 2.4 [0.96 to 3.7] | 2.5 [-0.69 to 4.3]

12. Secondary Outcome: Cognitive Function Measured by the Logical Memory, Recognition
Description: Pre-post difference in median category from baseline to 3 weeks on the Logical memory, recognition subscale. Scoring of this and all outcomes were based on best practices conveyed by study neuropsychologist during study design, and scoring approaches were chosen completely a priori. The recognition outcome of the LM test is derived from a series of conversions, as follows. First, the raw "process" score is converted to cumulative percentage (0-100). Because the cumulative percentage distribution is known to be skewed, best practice is to report scores as the following ordinal categorizations of cumulative percentages: <1, 3-9, 10-16, 17-25, 26-50, 51-75, and >75. To analyze them using simple statistics, these ordinal categories are converted to integer values (1-7), and the change in median ordinal category is presented along with 95% confidence intervals, generated by the Wilcoxon signed rank test with continuity correction.
Time Frame: baseline and 3 weeks
Population: No differences.
Measure: Median (95% Confidence Interval); unit: Ordinal category
Arm/Group | Low Insulin | Medium Insulin | High Insulin | Placebo
Number analyzed (Participants) | 6 | 7 | 9 | 6
Ordinal category | 1 [0 to 5] | 0 [0 to 2] | 0 [-1 to 2] | 1 [-1 to 3]

13. Secondary Outcome: Cognitive Function Measured by the Hopkins Verbal Learning Test - Revised (HVLT)
Description: as for outcome 7
Time Frame: baseline and 3 weeks
Measure: Mean (95% Confidence Interval); unit: T-score
Arm/Group | Low Insulin | Medium Insulin | High Insulin | Placebo
Number analyzed (Participants) | 6 | 7 | 9 | 6
T-score
  HVLT Immediate Recall | 3.0 [-5.0 to 11] | 1.6 [-5.8 to 9.0] | -4.6 [-11.1 to 2.0] | 0.0 [-8.0 to 8.0]
  HVLT Delayed Recall | -0.17 [-8.5 to 8.2] | 3.1 [-4.6 to 10.8] | -5.2 [-12.0 to 1.6] | 0.50 [-7.8 to 8.8]
  HVLT Recognition | 2.2 [-7.7 to 12.0] | -4.4 [-13.5 to 4.7] | -7.2 [-15.3 to 0.81] | 1.3 [-8.5 to 11.2]

14. Secondary Outcome: Cognitive Function Measured by the Visuospatial Memory Test - Revised (BVMT)
Description: as for outcome 7
Time Frame: 3 weeks
Measure: Mean (95% Confidence Interval); unit: T-scores
Arm/Group | Low Insulin | Medium Insulin | High Insulin | Placebo
Number analyzed (Participants) | 6 | 7 | 9 | 6
T-scores
  BVMT Immediate Recall | 5.5 [-23.2 to 13.2] | -8.6 [-15.7 to -1.4] | -3.0 [-9.3 to 3.3] | -11.8 [-19.6 to -4.1]
  BVMT Delayed Recall | -2.8 [-10.3 to 4.7] | -1.7 [-8.5 to 3.8] | -2.3 [-8.5 to 3.8] | -9.7 [-17.7 to -2.2]

15. Secondary Outcome: Cognitive Function Measured by the Stroop Color Word Test (CWT)
Description: as for outcome 7
Time Frame: baseline and 3 weeks
Measure: Mean (95% Confidence Interval); unit: T-score
Arm/Group | Low Insulin | Medium Insulin | High Insulin | Placebo
Number analyzed (Participants) | 6 | 7 | 9 | 6
T-score
  Word reading | -0.83 [-5.4 to 3.8] | 9.9 [5.6 to 14.4] | 2.8 [-0.97 to 6.5] | 1.7 [-2.9 to 6.3]
  Color naming | -2.3 [-6.7 to 2.0] | 6.3 [2.2 to 10.3] | 1.8 [-1.8 to 5.4] | 2.5 [-1.9 to 6.9]
  Color-word | 1.0 [-2.8 to 4.8] | 2.3 [-1.3 to 5.8] | -1.7 [-4.8 to 1.5] | 2.8 [-0.98 to 6.7]
  Interference | 2.2 [-1.8 to 6.2] | -2.9 [-6.6 to 0.85] | -1.8 [-5.1 to 1.5] | 1.3 [-2.7 to 5.3]

16. Secondary Outcome: Cognitive Function Measured by Fluency
Description: as for outcome 7
Time Frame: baseline and 3 weeks
Measure: Mean (95% Confidence Interval); unit: T-score
Arm/Group | Low Insulin | Medium Insulin | High Insulin | Placebo
Number analyzed (Participants) | 6 | 7 | 9 | 6
T-score
  Letter fluency | 4.7 [-1.3 to 10.6] | 5.0 [-0.53 to 10.5] | 2.9 [-2.0 to 7.8] | 1.3 [-4.6 to 7.3]
  Category fluency | 6.7 [0.12 to 13.2] | 4.7 [-1.4 to 10.8] | -1.8 [-7.1 to 3.6] | 1.5 [-5.1 to 8.1]

17. Secondary Outcome: Mood Measured by the Beck Depression Inventory - Second Edition
Description: Pre-post difference. Raw score. Range: 0-63. Higher score indicates more symptomatic.
Time Frame: baseline and 3 weeks
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Low Insulin | Medium Insulin | High Insulin | Placebo
Number analyzed (Participants) | 6 | 7 | 9 | 6
score on a scale | -2.5 [-5.5 to 0.49] | -2.3 [-5.1 to 0.48] | 0.22 [-2.2 to 2.7] | 1.3 [-2.6 to 5.3]

18. Secondary Outcome: Apathy Measured by the Apathy Scale
Description: Pre-post difference. Raw score. Range: 0-42. Higher score indicates more symptomatic.
Time Frame: baseline and 3 weeks
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Low Insulin | Medium Insulin | High Insulin | Placebo
Number analyzed (Participants) | 6 | 7 | 9 | 6
score on a scale | 0.67 [-3.3 to 4.6] | -0.86 [-4.5 to 2.8] | 1.7 [-1.6 to 4.9] | 1.3 [-2.6 to 5.3]

19. Secondary Outcome: Mood Measured by the Columbia Suicide Severity Rating (C-SSRS)
Description: Pre-post difference. Raw score. Range:1 or 0. 1 score - more symptomatic, 0 score - no symptoms.
Time Frame: baseline and 3 weeks
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Low Insulin | Medium Insulin | High Insulin | Placebo
Number analyzed (Participants) | 6 | 7 | 9 | 6
score on a scale | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]

20. Secondary Outcome: Motor Function as Measured by the United Parkinson's Disease Rating Scale (UPDRS-III)
Description: Pre-post difference. Raw score. Range: 0-72. Higher score indicates more symptomatic.
Time Frame: baseline and 3 weeks
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Low Insulin | Medium Insulin | High Insulin | Placebo
Number analyzed (Participants) | 6 | 7 | 9 | 6
score on a scale | -0.17 [-8.4 to 8.0] | 2.0 [-5.6 to 9.6] | -3.7 [-10.4 to 3.0] | -0.50 [-8.7 to 7.7]

21. Secondary Outcome: Cognitive Function Measured by Visuospatial Memory Test - Revised (BVMT Recognition)
Description: Pre-post difference in median category from baseline to 3 weeks on the Brief Visual Spatial Memory Test - Revised recognition. Scoring of this and all outcomes were based on best practices conveyed by study neuropsychologist during study design, and scoring approaches were chosen completely a priori. The recognition outcome of the BVMT test is derived from a series of conversions, as follows. First, the raw score is converted to cumulative percentage (0-100). Because the cumulative percentage distribution is known to be skewed, best practice is to report scores as the following ordinal categorizations of cumulative percentages: <2, 2-5, 6-10, 11-16, >16. To analyze them using simple statistics, these ordinal categories are converted to integer values (1-5), and the change in median ordinal category is presented along with 95% confidence intervals, generated by the Wilcoxon signed rank test with continuity correction.
Time Frame: baseline and 3 weeks
Measure: Median (95% Confidence Interval); unit: Ordinal category
Arm/Group | Low Insulin | Medium Insulin | High Insulin | Placebo
Number analyzed (Participants) | 6 | 7 | 9 | 6
Ordinal category | 0 [-3 to 1] | 0 [0 to 0] | 0 [-1 to 0] | -0.5 [-1 to 0]

ADVERSE EVENTS:
Time Frame: 5 weeks
Arm/Group | Low Insulin | Medium Insulin | High Insulin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/7 | 0/9 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/7 | 0/9 | 0/6
Other Adverse Events (participants affected / at risk) | 6/6 | 7/7 | 9/9 | 6/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low Insulin (N=6) | Medium Insulin (N=7) | High Insulin (N=9) | Placebo (N=6)
Nasal irritation (Skin and subcutaneous tissue disorders) | 4 (4) | 6 (11) | 6 (8) | 3 (3)
Muscle aches, pains, and sprains (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Respiratory/sinus symptoms (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0) | 4 (5) | 1 (1)
Falls (Ear and labyrinth disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (1)
Increased blood pressure (Blood and lymphatic system disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) — Increase deemed significant by PI
Nose bleeds (General disorders) | 3 (5) | 6 (9) | 6 (14) | 6 (8)
Other (General disorders) | 0 (0) | 5 (10) | 5 (5) | 2 (3) — Non significant laboratory results, dry eyes, sleeping issues, mood disorders, etc. All "other" AEs are categorized as "not related" or "probably not related" to study treatment
Headache (General disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Gastrointestinal issues (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Light-headedness, dizzyness (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-10-17): https://cdn.clinicaltrials.gov/large-docs/85/NCT04251585/Prot_SAP_000.pdf